CLINICAL TRIAL: NCT04207801
Title: A Phase II, Multicenter, Double-blind, Double-dummy, Placebo Controlled, Randomized, Study to Evaluate the Efficacy and Safety of Two Doses of AUR101 in Patients With Moderate-to-Severe Psoriasis
Brief Title: A Phase II Study to Evaluate Efficacy & Safety of AUR101 in Patients of Moderate-to-Severe Psoriasis
Acronym: INDUS-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aurigene Discovery Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUR101-201
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Chronic Plaque-type Psoriasis
Keywords: AUR101; Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm-1 400 mg BID (Experimental): 400 mg AUR101 twice daily
  Interventions: Drug: AUR101
- Arm-2 600 mg BID (Experimental): 600 mg AUR101 twice daily
  Interventions: Drug: AUR101
- Arm-3 - Matching Placebo BID (Placebo Comparator): Matching Placebo twice daily
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: AUR101 — Inhibitor of RORγ
  Other Names: No other names
  Arms: Arm-1 400 mg BID; Arm-2 600 mg BID
Drug: Matching Placebo — Drug-Placebo of AUR101 tablet
  Other Names: No other names
  Arms: Arm-3 - Matching Placebo BID

SUMMARY:
This will be a multicenter, double-blind, double-dummy, placebo controlled, randomized study to evaluate efficacy and safety of AUR101 (RORgamma inhibitor) in patients with moderate-to-severe psoriasis.

Approximately 90 patients with chronic moderate-to-severe plaque psoriasis will be randomized to the 2 dose groups of AUR101 and one group of Placebo. The patients will receive the treatment for 12 weeks.

DETAILED DESCRIPTION:
This will be a multicenter, double-blind, double-dummy, placebo controlled, randomized study to evaluate efficacy and safety of two doses of AUR101 in patients with moderate-to-severe psoriasis.

Approximately 90 patients with chronic moderate-to-severe plaque psoriasis (defined as Psoriasis Area and Severity Index (PASI) ≥12 and Body Surface Area (BSA) involved ≥10%) will be randomized to the 2 dose groups of AUR101 and placebo in the ratio of 1:1:1.

The patients in each arm will receive AUR101 of 400 mg twice daily or AUR101 600 mg twice daily or matching placebo twice daily for 12 weeks in a double blind, double dummy fashion.

Every patient will receive 12 weeks of treatment. All the patients will be followed up for 14 ± 2 days of their last dose for safety assessment.

A subset of approximately 25 patients, who consent, will be asked to come for plasma PK assessment in week 4 of dosing.

Efficacy evaluation will be done by PASI, DLQI and BSA assessment. Safety assessment will be done by AEs and regular lab assessment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Confirmed diagnosis of chronic plaque-type psoriasis, diagnosed at least 6 months before screening

  2. Psoriasis of at least moderate severity, defined as PASI≥12 and involved BSA≥10 % at screening and Day 1

  3. Adult males or females,≥18 to ≤ 65 years of age.

  4. Ability to communicate well with the investigator and to comply with the requirements of the entire study

  5. Willingness to give written informed consent (prior to any study related procedures being performed) and ability to adhere to the study restrictions and assessments schedule.

Exclusion Criteria:

* 1. History of erythrodermic, guttate, or pustular psoriasis within last 12 months

  2. Efficacy failure on any biologic (e.g. interleukin (IL) -17 antibodies or anti-TNF agents) for the treatment of psoriasis.

  3. Static 5-point IGA mod 2011 scale of 0 to 2 at screening or Day 1.

  4. BMI ≥ 35 kg/m2

  5. Current treatment or history of treatment for psoriasis with IL-17 or IL-12/23 antagonist biological agents within 6 months prior to study day 1

  6. Current treatment or history of treatment for psoriasis with other biological agents within 3 months prior to study day 1.

  7. Current treatment or history of treatment for psoriasis with non-biological systemic medications or phototherapy within 4 weeks prior to study day 1.

  8. Treatment with medicated topical agents within 2 weeks prior to study day 1.

  9. History or presence of any medical or psychiatric disease, or clinically significant laboratory at screening,

  10. Evidence of organ dysfunction

  11. Any major recent surgery history within 3 months prior to screening

  12. Alcohol abuse or drug abuse

  13. History of malignancy

  14. Positive for HIV, Hepatitis B or Hepatitis C at screening.

  15. Patient with known past history of systemic tuberculosis or currently suspected or known to have tuberculosis

  16. Patient expected to be started on anti-tubercular therapy either for treatment or prophylaxis of tuberculosis.

  17. Suspected tuberculosis infection as evident from a positive QuantiFERON TBGold test (QFT) at screening. Patients with a positive QFT test may participate in the study if further work up as per the opinion of the investigator .

  18. History of hypersensitivity or idiosyncratic reaction to any investigational RORgamma inhibitors or any of the excipients of study drug

  19. Past gastrointestinal surgery or recent (within 3 months) / current history of gastrointestinal disease.

  20. Positive pregnancy test for women of child bearing potential (WOCBP) at the screening or randomization visit

  21. Male patients with partners of childbearing potential not willing to use reliable contraception methods.

  22. Pregnant or lactating women or WOCBP who are neither surgically sterilized nor willing to use reliable contraceptive methods

  23. Has received another new chemical entity/investigational drug within 28 days or 5 half-lives of investigational drug prior to study day 1.

  24. Use of herbal remedies, mega dose vitamins and minerals during the 2 weeks prior to the first administration of investigational product.

  25. Patients who have received live or attenuated vaccine in the 4 weeks prior to study day 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shilendra Pandey, MSc, Study Chair — Aurigene Discovery Techologies Limited
Locations (9):
- India (9):
  - B.J Medical College & Civil Hospital, Ahmedabad, Gujarat
  - Kempegowda Institute of Medical Sciences, Bangalore, Karnataka
  - Sapthagiri Hospital, Bangalore, Karnataka
  - Triveni Polyclinic, Nagpur, Maharashtra
  - Shree Hospital and Critical Care Centre, Nagpur, Maharashtra
  - NKP Salve Institute of Medical Sciences and Lata Mangeshkar Hospital, Nagpur, Maharashtra
  - Sujata Birla Hospital & Medical Research Center, Nashik, Maharashtra
  - Apex Hospitals Private Limited, Jaipur, Rajasthan
  - Life Line Diagnostic Centre Cum Nursing Home, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: No
Not yet planned to share

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 90 patients were enrolled.. Out of these 90, 30 patients each were enrolled in 400 mg PO BID arm, 600 mg BID arm and placebo BID arm.
Groups:
- Arm-1: 400 mg AUR101 twice daily
  AUR101: Inhibitor of RORγ
- Arm-2: 600 mg AUR101 twice daily
  AUR101: Inhibitor of RORγ
- Arm-3: Matching Placebo twice daily
  Matching Placebo: Drug-Placebo of AUR101 tablet
Period: Overall Study
Arm/Group | Arm-1 | Arm-2 | Arm-3
Started | 30 | 30 | 30
Completed | 26 | 26 | 23
Not Completed | 4 | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm-1 | Arm-2 | Arm-3 | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 30 | 90
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (12.24) | 44.7 (9.72) | 44.4 (10.37) | 44.8 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 5 | 22
  Male | 21 | 22 | 25 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race is defined as "a category of humankind that shares certain distinctive physical traits." In this study, all pateints enrolled were of Indian descent
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 30 | 30 | 30 | 90
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0
    White | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  India | 30 | 30 | 30 | 90
Psoriasis Area and Severity Index (PASI) [Mean (Standard Deviation); unit: units on a scale] — PASI (Psoriasis Area and Severity Index) measures the intensity of redness, thickness, and scaling of the psoriasis is assessed as none (0), mild (1), moderate (2), severe (3), or very severe (4). The three intensity scores are added up for each of the four body regions to give subtotals A1, A2, A3, A4.
  Each subtotal is multiplied by the body surface area represented by that region. The percentage area affected by psoriasis is evaluated in the four regions of the body - Head and neck, Upper Limbs, Trunk and Lower Limbs.
  Minimum PASI Score is 0 and maximum is 72
  units on a scale | 26.1 (8.62) | 25.8 (10.7) | 24.2 (7.46) | 25.4 (8.97)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Achieving Psoriasis Area and Severity Index (PASI) 75 (i.e. 75% Reduction From Baseline PASI Score). (Scores Range From 0 (Minimum) to 30 (Maximum))
Description: Proportion of patients achieving Psoriasis Area and Severity Index (PASI) 75 (i.e. 75% reduction from baseline PASI score). (Scores range from 0 (minimum) to 30 (maximum)); The PASI is a scoring system to evaluate the baseline and response of therapy in psoriasis. Regulators commonly accept PASI 75 for measuring primary response of psoriasis in patients with Psoriasis. PASI 75 is a binary outcome that indicates a 75% or greater improvement in PASI from baseline
Time Frame: week 12
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm-1 | Arm-2 | Arm-3
Number analyzed (Participants) | 30 | 30 | 30
Participants | 18 | 19 | 8

2. Secondary Outcome: Proportion of Patients Achieving Psoriasis Area and Severity Index (PASI) 75 (i.e. 75% Reduction From Baseline PASI Score). (Scores Range From 0 (Minimum) to 30 (Maximum))
Description: Proportion of patients achieving Psoriasis Area and Severity Index (PASI) 75 (i.e. 75% reduction from baseline PASI score). (Scores range from 0 (minimum) to 30 (maximum)); The PASI is a scoring system to evaluate the baseline and response of therapy in psoriasis. PASI 75 is a binary outcome that indicates a 75% or greater improvement in PASI from baseline. These secondary measures are measured as Week 4 and Week 8 from the initiation of study drug therapy.
Time Frame: Week 4 and Week 8 from study drug initiation for these secondary outcomes measures
Population: PASI-75 Response at Week 8 for ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm-1 | Arm-2 | Arm-3
Number analyzed (Participants) | 30 | 30 | 30
Participants
  PASI-75 Response at Week 8 | 10 | 4 | 5
  PASI-75 Response at Week 4 | 1 | 1 | 0

3. Secondary Outcome: Proportion of Patients Achieving Psoriasis Area and Severity Index (PASI) 50 (i.e. 50% Reduction From Baseline PASI Score). (Scores Range From 0 (Minimum) to 30 (Maximum))
Description: Proportion of patients achieving Psoriasis Area and Severity Index (PASI) 50 (i.e. 50% reduction from baseline PASI score). (Scores range from 0 (minimum) to 30 (maximum)); The PASI is a scoring system to evaluate baseline and response of therapy in psoriasis. Like PASI 75, the PASI-50 is a binary outcome that indicates a 50% or greater improvement in PASI from baseline. PASI-50 is measured at Week 4, Week 8 and Week 12, as part of this secondary outcome measure.
Time Frame: Week 4, Week 8 and Week 12
Population: PASI-50 at week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Arm-1 | Arm-2 | Arm-3
Number analyzed (Participants) | 30 | 30 | 30
Participants
  PASI-50 at Week 12 | 23 | 20 | 14
  PASI-50 at Week 8 | 16 | 13 | 10
  PASI-50 at Week 4 | 10 | 3 | 3

4. Secondary Outcome: Proportion of Patients Achieving Investigator Global Assessment (IGA) Score of 0 or 1
Description: The proportion of patients achieving Investigator Global Assessment (IGA) score of 0 or 1 (Scores range from 0 (0 or 1 clear to mild) to 4 (severe)); The 5-point IGA has a more stringent definition for a score of 1 ("almost clear"); This secondary measure is measured at Week 4, Week 8 and Week 12. The sponsor has represented the proportion in % form by multiplying by 100. The sponsor has done that in CSR (Clinical Study Report) as well
Time Frame: Week 4, Week 8 and Week 12
Population: ITT (Intention to Treat) population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm-1 | Arm-2 | Arm-3
Number analyzed (Participants) | 30 | 30 | 30
Participants
  IGA Response of 0 or 1 at Week 12 | 17 | 16 | 8
  IGA Response of 0 or 1 at Week 8 | 7 | 4 | 2
  IGA Response of 0 or 1 at Week 4 | 0 | 0 | 0

5. Secondary Outcome: Percent Change From Baseline in Psoriasis Area and Severity Index (PASI) Score.
Description: The Psoriasis Area Severity Index (PASI) is an index used to express the severity of psoriasis. It combines the severity (erythema, induration and desquamation) and percentage of affected area. Percent change from baseline in Psoriasis Area and Severity Index (PASI) score. The PASI is a widely used instrument in psoriasis trials that assesses and grades the severity of psoriatic lesions and the patient's response to treatment. It produces a numeric score ranging from 0 to 72. This outcome measures the percentage decrease in PASI from baseline at various pre-specified timepoints
Time Frame: week 4,8 and 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Percent change from baseline in PASI
Arm/Group | Arm-1 | Arm-2 | Arm-3
Number analyzed (Participants) | 30 | 30 | 30
Percent change from baseline in PASI
  Percent Change in PASI at week12 | -68.1 (33.68) | -60.3 (43.04) | -43.8 (36.19)
  Percent Change in PASI at week 8 | -52.4 (33.68) | -39.9 (39.36) | -32.6 (40.13)
  Percent Change in PASI at week 4 | -28.2 (27.84) | -20.4 (26.76) | -15.5 (20.35)

6. Secondary Outcome: Change From Baseline in Investigator Global Assessment (IGA) Scale
Description: The 5-point IGA has a more stringent definition for a score of 1 ("almost clear") compared with 6-point IGA/Physician's Global Assessment (PGA) tools used in previous trials of other biologics in moderate-to-severe psoriasis. The IGA 0/1 rate is considered robust, demonstrating a strong association with PASI 90. The results for the 5-point IGA are expected to show the same association. This endpoint measures the percent change from baseline in Investigator Global Assessment (IGA) scale (Scores range from 0 (0 or 1 clear to mild) to 4 (severe)) at pre-specified time points.
Time Frame: week 4,8 and 12
Population: ITT population
Measure: Mean (Standard Deviation); unit: % decrease in IGA score
Arm/Group | Arm-1 | Arm-2 | Arm-3
Number analyzed (Participants) | 30 | 30 | 30
% decrease in IGA score
  Percent Change from baseline in IGA at week 12 | -50.8 (31.74) | -46.9 (36.72) | -28.9 (29.18)
  Percent Change from baseline in IGA at week 8 | -34.2 (24.4) | -24.4 (27.15) | -19.4 (19.74)
  Percent Change from baseline in IGA at week 4 | -12.5 (18.41) | -8.9 (15.46) | -3.1 (9.41)

7. Secondary Outcome: Change From Baseline to Week 4, 8 and 12 in Percent Body Surface Area (BSA) Involved
Description: BSA assessment measures the total area of the body affected by psoriasis. The body surface area (BSA) of involvement is an important indicator during the evaluation of psoriasis severity. In this secondary outcome measure, the change from baseline to week 4, 8 and 12 in percent Body Surface Area (BSA) involved is measured
Time Frame: week 4,8 and 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: % decrease in BSA (Body Surface Area)
Arm/Group | Arm-1 | Arm-2 | Arm-3
Number analyzed (Participants) | 30 | 30 | 30
% decrease in BSA (Body Surface Area)
  BSA% change at Week 12 | -57.6 (35.03) | -56.1 (39.65) | -29.9 (34.33)
  BSA % Change at Week 8 | -35.3 (30.57) | -30.2 (35.15) | -20.4 (32.89)
  BSA % Change at Week 4 | -8.3 (19.18) | -10.0 (20.28) | -8.8 (17.72)

8. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI)
Description: The DLQI is a validated, 10-question, self-reported questionnaire to evaluate the patient's perception of the impact of psoriasis on their quality of life. The DLQI Scores range from 0 to 30, and higher scores indicate greater health-related quality-of-life impairment.
  The DLQI questionnaire is divided into 6 commonly identified categories and is rated on a 4-point scale. This secondary outcome measures the change from baseline to week 4, 8 and 12 in Dermatology Life Quality Index (DLQI) score. The minimum value is 0 and maximum is 4
Time Frame: Week 4,8 and 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Percent change from baseline in DLQI
Arm/Group | Arm-1 | Arm-2 | Arm-3
Number analyzed (Participants) | 30 | 30 | 30
Percent change from baseline in DLQI
  Percent Change from Baseline in DLQI score at week 12 | -47.1 (89.45) | -49.1 (47.53) | -32.7 (49.46)
  Percent Change from Baseline in DLQI score at week 8 | -31.9 (89.83) | 33.0 (46.9) | -25.6 (48.36)
  Percent Change from Baseline in DLQI score at week 4 | -9.9 (82.47) | -16.9 (48.94) | -14.1 (33.16)
Statistical Analysis 1: Comparison: Arm-1 vs Arm-2 vs Arm-3; Efficacy of AUR101 was tested against placebo with respect to the primary endpoint (PASI75 response). A sample size of 25 in each of the three arms provided an 80% power with a one-sided Type I error of 0.05, if the true placebo response rate was 7% and the response rate on investigational arm(s) was 35%. The sample size was increased to 30 to account for ~ 15-20% dropouts over the study period; Test type: Superiority; p = 0.01, Fisher Exact

ADVERSE EVENTS:
Time Frame: From enrolment to 2 week follow up
Description: No difference
Arm/Group | Arm-1 | Arm-2 | Arm-3
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 2/30
Other Adverse Events (participants affected / at risk) | 2/30 | 3/30 | 1/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm-1 (N=30) | Arm-2 (N=30) | Arm-3 (N=30)
COVID-19 Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Psoriatic Erythroderma (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm-1 (N=30) | Arm-2 (N=30) | Arm-3 (N=30)
Pruritus (General disorders) | 2 (2) | 1 (1) | 1 (1)
Depressed Mood (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT04207801/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/01/NCT04207801/SAP_001.pdf